CLINICAL TRIAL: NCT03207620
Title: Interrelation Between Bronchial Asthma and Smoking
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Abd El-gayed Eid, principal investigator, Assiut University
Other Study IDs: IBBAAS
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum and serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smoker asthmatics: * Asthma control questionnaire (ACQ) score
  * Spirometry
  * Sputum cytology
  Interventions: Diagnostic Test: using serum periostin and eotaxin-2 level; Diagnostic Test: airway corticosteroid sensitivity
- non-smoker asthmatics: * Asthma control questionnaire (ACQ) score
  * Spirometry
  * Sputum cytology
  Interventions: Diagnostic Test: using serum periostin and eotaxin-2 level; Diagnostic Test: airway corticosteroid sensitivity

INTERVENTIONS:
Diagnostic Test: using serum periostin and eotaxin-2 level — collect serum sample from each group and detection of serum periostin and eotaxin-2 are using Eliza kits.
  each group is divided into two groups (patients who are already using ICS and patients who do not use ICS) and we compare between to groups in airway hypersensitivity.
Diagnostic Test: airway corticosteroid sensitivity — each group is divided into two groups (patients who are already using inhaled corticosteroid ICS and patients who do not use ICS) and we compare between to groups in airway hypersensitivity.

SUMMARY:
Smoking occurs frequently in patients with asthma. Recent surveys on smoking prevalence report 21-26% current smokers in populations of patients with asthma. Detrimental effects of active smoking in asthma include worse asthma control, an impaired response to corticosteroids and accelerated lung function decline.

DETAILED DESCRIPTION:
The mechanisms by which cigarette smoking contributes to disease severity in asthma are incompletely understood, but it has been suggested that cigarette smoking may change inflammation and airway remodelling in asthma to become more similar to that in COPD (chronic obstructive pulmonary disease).

Any form of tobacco use, especially cigarette smoking, plays an important role in this disease. Asthmatic smokers are prone to several negative outcomes. Cigarette smoking by itself is associated with airway inflammation and features of airway remodelling including increased epithelial proliferation, squamous cell metaplasia, goblet cell hyperplasia, smooth muscle hypertrophy, and increases in bronchial glands mass.

Corticosteroid insensitivity is an important clinical feature of asthma, particularly in patients with severe disease and smokers. The mechanisms of corticosteroid insensitivity in asthmatic patients are poorly understood.

One of the major problems in the treatment of smoking asthma patients is the lack of efficacy data in this group of patients as smokers have almost always been excluded from studies on asthma due to perceived concerns about recruiting patients with COPD. Therefore, there is a lack of specific information about the treatment of asthma in smokers. The asthmatic smoker is a special phenotype with important therapeutic and prognostic clinical implications.

ELIGIBILITY:
Inclusion criteria:

1. Stable asthmatic patients (however smokers, or non-smokers) will be included (stable asthmatic defined as no emergency clinic or hospital visit, oral corticosteroid prescription, or change in asthma treatment in the past month) and (Current smoking was defined as 5 or more cigarettes per day and a smoking history of 5 pack years or greater).
2. Treatment with long-acting b2-agonists, and leukotriene receptor antagonists was allowed.

Exclusion criteria:

1. Acute severe asthma.
2. Causes of airway obstruction other than asthma as COPD patients, bronchiectasis……etc.
3. Age <18 and >45 years old.
4. Body mass index >35.
5. Requirement for treatment with or the presence of conditions likely to be exacerbated by oral corticosteroids
6. The intention to stop smoking. Eligibility for the study required demonstration of reversible airflow obstruction (FEV1 bronchodilator response to b2 agonist of >12% [and >200 mL]) or a positive methacholine test result. All lung function assessments met relevant international consensus guidelines.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Stable asthmatic patients (however smokers, or non-smokers) will be included (stable asthmatic defined as no emergency clinic or hospital visit, oral corticosteroid prescription, or change in asthma treatment in the past month) and (Current smoking was defined as 5 or more cigarettes per day and a smoking history of 5 pack years or greater).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
serum periostin | one day
  detect its level in serum
Serum eotaxin-2 | One day
  detect its level in serum

SECONDARY OUTCOMES:
Spirometry | one day
  pre- and post bronchodilator FEV1 will be measured.
Sputum cytology | one day
  detect proportion of eosinophils and neutrophils in sputum cytology.
airway corticosteroid sensitivity | one month
  Airway corticosteroid sensitivity will be assessed by change in pre-bronchodilator FEV1 (forced expiratory volume at one second) .

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Eid, master, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vozoris NT, Stanbrook MB. Smoking prevalence, behaviours, and cessation among individuals with COPD or asthma. Respir Med. 2011 Mar;105(3):477-84. doi: 10.1016/j.rmed.2010.08.011. Epub 2010 Sep 17. PMID 20850288
- [Background] Cerveri I, Cazzoletti L, Corsico AG, Marcon A, Niniano R, Grosso A, Ronzoni V, Accordini S, Janson C, Pin I, Siroux V, de Marco R. The impact of cigarette smoking on asthma: a population-based international cohort study. Int Arch Allergy Immunol. 2012;158(2):175-83. doi: 10.1159/000330900. Epub 2012 Jan 26. PMID 22286571
- [Background] Chaudhuri R, McSharry C, McCoard A, Livingston E, Hothersall E, Spears M, Lafferty J, Thomson NC. Role of symptoms and lung function in determining asthma control in smokers with asthma. Allergy. 2008 Jan;63(1):132-5. doi: 10.1111/j.1398-9995.2007.01538.x. PMID 18053022
- [Background] Clatworthy J, Price D, Ryan D, Haughney J, Horne R. The value of self-report assessment of adherence, rhinitis and smoking in relation to asthma control. Prim Care Respir J. 2009 Dec;18(4):300-5. doi: 10.4104/pcrj.2009.00037. PMID 19562233
- [Background] Chalmers GW, Macleod KJ, Little SA, Thomson LJ, McSharry CP, Thomson NC. Influence of cigarette smoking on inhaled corticosteroid treatment in mild asthma. Thorax. 2002 Mar;57(3):226-30. doi: 10.1136/thorax.57.3.226. PMID 11867826
- [Background] Lazarus SC, Chinchilli VM, Rollings NJ, Boushey HA, Cherniack R, Craig TJ, Deykin A, DiMango E, Fish JE, Ford JG, Israel E, Kiley J, Kraft M, Lemanske RF Jr, Leone FT, Martin RJ, Pesola GR, Peters SP, Sorkness CA, Szefler SJ, Wechsler ME, Fahy JV; National Heart Lung and Blood Institute's Asthma Clinical Research Network. Smoking affects response to inhaled corticosteroids or leukotriene receptor antagonists in asthma. Am J Respir Crit Care Med. 2007 Apr 15;175(8):783-90. doi: 10.1164/rccm.200511-1746OC. Epub 2007 Jan 4. PMID 17204725
- [Background] James AL, Palmer LJ, Kicic E, Maxwell PS, Lagan SE, Ryan GF, Musk AW. Decline in lung function in the Busselton Health Study: the effects of asthma and cigarette smoking. Am J Respir Crit Care Med. 2005 Jan 15;171(2):109-14. doi: 10.1164/rccm.200402-230OC. Epub 2004 Oct 14. PMID 15486340
- [Background] Lange P, Scharling H, Ulrik CS, Vestbo J. Inhaled corticosteroids and decline of lung function in community residents with asthma. Thorax. 2006 Feb;61(2):100-4. doi: 10.1136/thx.2004.037978. PMID 16443705
- [Background] O'Byrne PM, Lamm CJ, Busse WW, Tan WC, Pedersen S; START Investigators Group. The effects of inhaled budesonide on lung function in smokers and nonsmokers with mild persistent asthma. Chest. 2009 Dec;136(6):1514-1520. doi: 10.1378/chest.09-1049. Epub 2009 Aug 26. PMID 19710291
- [Background] Tamimi A, Serdarevic D, Hanania NA. The effects of cigarette smoke on airway inflammation in asthma and COPD: therapeutic implications. Respir Med. 2012 Mar;106(3):319-28. doi: 10.1016/j.rmed.2011.11.003. Epub 2011 Dec 22. PMID 22196881
- [Background] Chatkin JM, Dullius CR. The management of asthmatic smokers. Asthma Res Pract. 2016 Jun 20;2:10. doi: 10.1186/s40733-016-0025-7. eCollection 2016. PMID 27965778
- [Background] Hiroshima K, Iyoda A, Shibuya K, Hoshino H, Haga Y, Toyozaki T, Shiba M, Baba M, Fujisawa T, Ohwada H. Evidence of neoangiogenesis and an increase in the number of proliferating cells within the bronchial epithelium of smokers. Cancer. 2002 Oct 1;95(7):1539-45. doi: 10.1002/cncr.10850. PMID 12237923
- [Background] Mathe G, Santelli G, Gouveia J, Lemaigre G, Misset JL, Gros F, Homasson JP, Kim B, Sudre MC, Gaget H. Correlation of bronchial epidermoid metaplasia with level of tobacco consumption in heavy smokers. Cancer Detect Prev. 1986;9(1-2):79-81. PMID 3731197
- [Background] Niewoehner DE, Kleinerman J, Rice DB. Pathologic changes in the peripheral airways of young cigarette smokers. N Engl J Med. 1974 Oct 10;291(15):755-8. doi: 10.1056/NEJM197410102911503. No abstract available. PMID 4414996
- [Background] Cosio MG, Hale KA, Niewoehner DE. Morphologic and morphometric effects of prolonged cigarette smoking on the small airways. Am Rev Respir Dis. 1980 Aug;122(2):265-21. doi: 10.1164/arrd.1980.122.2.265. PMID 7416603
- [Background] McSharry C, Spears M, Chaudhuri R, Cameron EJ, Husi H, Thomson NC. Increased sputum endotoxin levels are associated with an impaired lung function response to oral steroids in asthmatic patients. J Allergy Clin Immunol. 2014 Nov;134(5):1068-75. doi: 10.1016/j.jaci.2014.08.022. Epub 2014 Sep 26. PMID 25262463
- [Background] Decramer M, Louis R, Joos G, De Vuyst P, Mast B, Mehuys A; Pulmonary Advisory Board. (Ex-)smoking asthma patients in general and specialized Belgian practice. Respir Med. 2011 Aug;105(8):1203-10. doi: 10.1016/j.rmed.2011.02.017. Epub 2011 Mar 16. PMID 21414762